CLINICAL TRIAL: NCT01730456
Title: A MULTICENTER, OPEN-LABEL, SINGLE ARM, LONG TERM EXTENSION STUDY OF WA19926 TO DESCRIBE SAFETY DURING TREATMENT WITH TOCILIZUMAB IN PATIENTS WITH EARLY, MODERATE TO SEVERE RHEUMATOID ARTHRITIS
Brief Title: A Long-Term Extension Study of RoActemra/Actemra (Tocilizumab) in Patients With Early Moderate to Severe Rheumatoid Arthritis Who Completed Study WA19926
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML28133
Record Dates: First submitted 2012-11-15; First posted 2012-11-21 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tocilizumab

ARMS (1):
- RoActemra/Actemra (Experimental)
  Interventions: Drug: tocilizumab [RoActemra/Actemra]

INTERVENTIONS:
Drug: tocilizumab [RoActemra/Actemra] — 8 mg/kg iv every 4 weeks, up to 104 weeks

SUMMARY:
This multicenter, open-label, single arm, long-term extension study will evaluate the safety and efficacy of RoActemra/Actemra (tocilizumab) in patients with early moderate to severe rheumatoid arthritis who completed the WA19926 core study. Patients will receive RoActemra/Actemra 8 mg/kg intravenously every 4 weeks for up to 104 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/= 18 years of age
* Patients who complete their last WA19926 core study visit (Week 104) and who may benefit from study drug treatment according to the Investigator's assessment
* No current or recent adverse event or laboratory finding preventing the use of the study drug dose of RoActemra/Actemra 8 mg/kg at baseline visit
* Receiving treatment on an outpatient basis
* Females of childbearing potential must agree to use at least one adequate method of contraception, including a method with a failure rate of <1% per year, during the treatment period

Exclusion Criteria:

* Pregnant or lactating women
* Patients who have prematurely withdrawn from the WA19926 core study for any reason
* Treatment with an investigational agent or cell-depleting therapies since the last administration of study drug in the WA19926 core study
* Immunization with a live/attenuated vaccine since the last administration of study drug in the WA19926 core study
* Diagnosis since last WA19926 visit (Week 104) of rheumatic autoimmune disease other than rheumatoid arthritis
* Diagnosis since last WA19926 visit (Week 104) of inflammatory joint disease other than rheumatoid arthritis
* Inadequate liver, hematologic or renal function
* History of severe allergic or anaphylactic reactions to humanized or murine monoclonal antibodies
* Known active or history of recurrent infections
* Evidence of active malignant disease, malignancies within the previous 10 years (except for basal cell carcinoma of the skin that has been excised and cured), or breast cancer diagnosed within the previous 20 years
* Uncontrolled disease states, such as asthma or inflammatory bowel disease, where flares are commonly treated with oral or parenteral corticosteroids

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2012-10; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Long-term safety: Incidence of adverse events | approximately 3 years

SECONDARY OUTCOMES:
Change in disease activity: Disease Activity Score 28 - erythrocyte sedimentation rate (DAS28-ESR) and/or Simplified Disease Activity Index (SDAI) | from baseline to Week 104
Change in total tender joint count (TJC) / swollen joint count (SJC) | from baseline to Week 104
Proportion of patients achieving sustained drug-free remission, defined as clinical remission based on DAS28-ESR <2.6 and/or SDAI </=3 for two consecutive visits (every 12 weeks) followed by RoActemra/Actemra discontinuation after the 2nd visit | approximately 3 years
Time to rheumatoid arthritis flare in patients who have entered drug-free remission | approximately 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Skopje, North Macedonia